CLINICAL TRIAL: NCT04471857
Title: Using Medical Hypnotherapy in Children With Defecation Disorders
Brief Title: Hypnosis for Children Undergoing Anorectal Manometry
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 recruitement stopped since intended sample size was an estimation and not based on power calculation
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Frederick Woodley, PhD, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB15-00864
Record Dates: First submitted 2020-06-30; First posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Constipation
Keywords: hypnosis; anorectal manometry; child
MeSH Terms: conditions — Constipation | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A blinded observer assessed child distress during anorectal manometry
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis (Experimental): A brief session of hypnosis just before child starts with anorectal manometry
  Interventions: Behavioral: Hypnosis
- Control (No Intervention): No hypnosis session, standard care

INTERVENTIONS:
Behavioral: Hypnosis
  Arms: Hypnosis

SUMMARY:
Partially blinded randomized controlled trial investigating the effect of a brief session of hypnosis prior to anorectal manometry in children

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-18 who are scheduled to undergo anorectal manometry testinf.
* ASA classification I to II.
* Both parents and children have sufficient English language proficiency.
* Both parents and children are willing to fill out the questionnaires involved in this study.

Exclusion Criteria:

* ASA classification III, IV (children with a chronic or severe disease).
* Children with a metabolic, endocrine or neuromuscular disorder or mental illness.
* Children with anorectal malformations or previous anorectal surgery.
* Children with developmental delay
* Children with diagnosed emotional or behavioral disorders

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this study will be the assessment of distress as measured by the non-blinded observer. | Periprocedural
  The non-blinded observer will use the Observation Scale of Behavioral Distress (OSBD) to assess the periprocedural distress of the child. The OSBD records the presence or absence of thirteen operationally-defined behaviors, which indicate discomfort (e.g. cry, verbal resistance, information seeking) at 15-second intervals throughout the procedure. The behaviors are given a score ranging from 1 to 4 according to the severity of distress that is expressed by that behavior. The recorded score during a 15-second interval can range from zero (no distress) to 33.5 (extreme distress). The total scores will be summed up and then divided by the number of 15-second intervals to obtain a mean distress score.

SECONDARY OUTCOMES:
Periprocedural distress as measured by the blinded observer | Periprocedural
  The blinded observer rates the child's distress on a 4-point Likert scale ranging from 0 (not anxious at all) to 3 (extremely anxious). Ratings are based on facial features, crying, and physical movements. The blinded observer reports the highest (i.e. peak), most common (i.e. typical),and the lowest level of distress. We will compare the highest and most common levels of distress between groups, as we believed these levels of distress are most clinically relevant.
Child-reported levels of distress | Right after anorectal manometry (same day)
  The child will be asked to rate the amount of distress experienced (unpleasantness, nervousness, and anxiety) during the manometry on a 5-point Likert scale ranging from 0 (not at all) to 4 (very much). They are also asked to rate the pain of the procedure on an analogous scale of 0 (no pain) to 10 (extremely painful). Children who received hypnosis are asked if they believed that it helped them to relax on a 5-point Likert scale ranging from 0 (not at all) to 4 (very much).
Parent-reported levels of distress | Right after anorectal manometry (same day)
  The parent accompanying the child will be asked to rate the amount of distress of the child (unpleasantness, nervousness, and anxiety) during the manometry on a 5-point Likert scale ranging from 0 (not at all) to 4 (very much). They are also asked to rate the pain of the procedure on an analogous scale of 0 (no pain) to 10 (extremely painful). Parents of children who received hypnosis are asked if they believed that it helped the child to relax on a 5-point Likert scale ranging from 0 (not at all) to 4 (very much).
Difficulty of procedure | Right after anorectal manometry (same day)
  The motility nurse will report if all parts of the procedure could be performed properly and rates the degree of difficulty of the procedure on a 5-point Likert scale ranging from 0 (not at all) to 4 (very much).
Difficulty of hypnosis | Right after anorectal manometry (same day)
  The hypnotherapist rates the degree of difficulty of the hypnosis on a similar 5-point Likert scale ranging from 0 (not at all) to 4 (very much).
Manometry outcomes | Periprocedural
  Procedural outcomes of the children undergoing anorectal manometry will be recorded and compared between groups. This includes: resting pressure, squeeze pressure, squeeze duration, push test, duration of procedure.

IPD SHARING:
Plan to Share IPD: No